CLINICAL TRIAL: NCT03291314
Title: Phase II Clinical Trial on the Combination of Avelumab and Axitinib for the Treatment of Patients With Recurrent Glioblastoma
Brief Title: Clinical Trial on the Combination of Avelumab and Axitinib for the Treatment of Patients With Recurrent Glioblastoma
Acronym: GliAvAx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Bart Neyns, Prof. Dr., Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-BN-001
Record Dates: First submitted 2017-06-29; First posted 2017-09-25 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Recurrent Glioblastoma (WHO-Grade IV Glioma)
MeSH Terms: conditions — Glioblastoma | interventions — Axitinib; avelumab

STUDY DESIGN:
Intervention Model Description: Open label, single-center, stratified phase II clinical trial.
  Patients will be stratified according to their baseline use of corticosteroids: <Stratum A> = no need for corticosteroids and <Stratum B> = baseline need for steroid treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Axitinib + Avelumab (Experimental): On day 1 of the treatment phase, patients recruited to this arm will initiate concomitant continuous daily treatment with axitinib (InlytaTM, 5 mg comp BID) in combination with avelumab (10 mg/kg IV Q2 weeks)
  Interventions: Drug: Axitinib; Drug: Avelumab
- Axitinib (+Avelumab) (Experimental): On day 1 of the treatment phase, patients recruited to this arm will initiate treatment with continuous daily axitinib (InlytaTM, 5 mg comp BID).
  Patients who tolerate treatment with axitinib and are able to taper the dose of corticosteroids to a maximal daily dose of 8 mg methylprednisolone (or an equivalent dose of another oral corticosteroid) will initiate combination therapy with avelumab (10 mg/kg IV Q2 weeks) on day 43, following the the first MRI-based tumor response evaluation in week 6.
  Patients who do not tolerate monotherapy with axitinib, or cannot decrease their daily dose of corticosteroids to a maximal daily dose of 8 mg methylprednisolone will not be allowed to initiate avelumab treatment.
  Interventions: Drug: Axitinib; Drug: Avelumab

INTERVENTIONS:
Drug: Axitinib — 1. Axitinib, a VEGFR-specific small molecule tyrosine kinase inhibitor (Tki) has demonstrated anti-tumor activity when evaluated as a mono-therapy and in combination with lomustine for the treatment of patients with recGB (EudraCT 2011-000900-16) [7].
  Other Names: InlytaTM
Drug: Avelumab — 2. Avelumab (MSB00107; anti-PD-L1) is a fully human anti-PD-L1 IgG1 monoclonal antibody (mAb) that has demonstrated anti-tumor activity in several tumor types.
  Other Names: MSB00107

SUMMARY:
Phase II clinical trial on the combination of avelumab and axitinib for the treatment of patients with recurrent glioblastoma (histologically confirmed WHO grade IV glioma), at documented recurrence/progression following prior treatment with surgery, radiation therapy and temozolomide.

DETAILED DESCRIPTION:
High-grade gliomas of the central nervous system (CNS) are characterized by profound tumor related neo-angiogenesis, and intracranial perilesional edema. Glioblastoma (WHO-grade IV glioma) expresses high levels of VEGF and frequently carries an amplified gene copy numbers of the VEGFR2, KIT and PDGFR or EGFR genes, key mediators of the process of cancer related neo-angiogenesis. In patient diagnosed with recurrence/progression glioblastoma (recGB) following prior therapy with surgery, radiation therapy and temozolomide, cytotoxic salvage therapies resulted in a best overall response rate of 5 to 10%, 6-month PFS rates of 9% to 21%, and a median OS of 25 to 30 weeks. No treatment option has demonstrated to improve the survival expectancy of recGB patients in a randomized clinical trial. Bevacizumab treatment has been registered by FDA based on objective tumor response rates and PFS results obtained in uncontrolled phase II trials. There is currently no treatment registered by EMA for the indication of recGB.

Axitinib, a VEGFR-specific small molecule tyrosine kinase inhibitor (Tki) has demonstrated anti-tumor activity when evaluated as a mono-therapy and in combination with lomustine for the treatment of patients with recGB (EudraCT 2011-000900-16). Immunocytochemical profiling of the peripheral blood of recurrent GBM patients treated with axitinib or axitinib plus lomustine showed that axitinib treatment increases the number of naive CD8+ T cells and central memory CD4+ and CD8+ T cells. There was also a reduction of TIM3 expression and an increased cytokine production in the patients treated with axitinib. Upon progression during axitinib treatment patients displayed an increased immune suppression with an increased number of Treg, an increased PD-1 expression on CD4+ and CD8+ T cells, and a reduced T cell functionality.

Avelumab (MSB00107; anti-PD-L1) is a fully human anti-PD-L1 IgG1 monoclonal antibody (mAb) that has demonstrated anti-tumor activity in several tumor types. Expression of PD-L1 by tumor cells has been correlated with a higher probability for respons to avelumab throughout different tumor types. Glioblastoma has been reported to expresses the PD-L1 ligand.

In preclinical mouse models we demonstrated that axitinib reduces the immune suppressive microenvironment through reduction of the suppressive capacity of monocytic MDSCs (both in intra-cranial as well as subcutaneous tumors). Moreover, it also increased the number of tumor-infiltrating T cells. When we combined axitinib with active immunotherapy in the form of CTLA4 blockade not only a supplementary reduction of the suppressive capacity of these monocytic MDSCs was found, but also a reduction of the intratumoral granulocytic MDSCs and an increased antigen-presenting function of intratumoral DCs (manuscript accepted for publication in High-grade gliomas of the central nervous system (CNS) are characterized by profound tumor related neo-angiogenesis, and intracranial perilesional edema. Glioblastoma (WHO-grade IV glioma) expresses high levels of VEGF and frequently carries an amplified gene copy numbers of the VEGFR2, KIT and PDGFR or EGFR genes, key mediators of the process of cancer related neo-angiogenesis. In patient diagnosed with recurrence/progression glioblastoma (recGB) following prior therapy with surgery, radiation therapy and temozolomide, cytotoxic salvage therapies resulted in a best overall response rate of 5 to 10%, 6-month PFS rates of 9% to 21%, and a median OS of 25 to 30 weeks. No treatment option has demonstrated to improve the survival expectancy of recGB patients in a randomized clinical trial. Bevacizumab treatment has been registered by FDA based on objective tumor response rates and PFS results obtained in uncontrolled phase II trials. There is currently no treatment registered by EMA for the indication of recGB.

Axitinib, a VEGFR-specific small molecule tyrosine kinase inhibitor (Tki) has demonstrated anti-tumor activity when evaluated as a mono-therapy and in combination with lomustine for the treatment of patients with recGB (EudraCT 2011-000900-16). Immunocytochemical profiling of the peripheral blood of recurrent GBM patients treated with axitinib or axitinib plus lomustine showed that axitinib treatment increases the number of naive CD8+ T cells and central memory CD4+ and CD8+ T cells. There was also a reduction of TIM3 expression and an increased cytokine production in the patients treated with axitinib. Upon progression during axitinib treatment patients displayed an increased immune suppression with an increased number of Treg, an increased PD-1 expression on CD4+ and CD8+ T cells, and a reduced T cell functionality.

Avelumab (MSB00107; anti-PD-L1) is a fully human anti-PD-L1 IgG1 monoclonal antibody (mAb) that has demonstrated anti-tumor activity in several tumor types. Expression of PD-L1 by tumor cells has been correlated with a higher probability for respons to avelumab throughout different tumor types. Glioblastoma has been reported to expresses the PD-L1 ligand.

In preclinical mouse models we demonstrated that axitinib reduces the immune suppressive microenvironment through reduction of the suppressive capacity of monocytic MDSCs (both in intra-cranial as well as subcutaneous tumors). Moreover, it also increased the number of tumor-infiltrating T cells. When we combined axitinib with active immunotherapy in the form of CTLA4 blockade not only a supplementary reduction of the suppressive capacity of these monocytic MDSCs was found, but also a reduction of the intratumoral granulocytic MDSCs and an increased antigen-presenting function of intratumoral DCs (manuscript accepted for publication in American Journal of Cancer Research).

The rational for combining avelumab with for the treatment of recGB is based on the potential of axitinib to normalize the glioblastoma associated neo-vasculature, counteracting the immunosuppressive role of VEGF in the tumor microenvironment and controlling intracranial edema. These features may result in a synergistic anti-tumor effect with the PD-L1 inhibitory mAb avelumab. In addition, axitinib may reduce the inflammatory edema related to the anti-tumor effect mediated by PD-L1 inhibition with avelumab.

Patients with recGBM often develop neurological symptoms related to perilesional edema. Corticosteroids are considered a standard of care for controlling intracranial edema in patients with glioblastoma. High dose corticosteroids however are known to be immunosuppressive and are likely to counteract the therapeutic effect of anti-PD-L1 antibody therapy. Axitinib has the capacity to control recGBM associated edema of the brain. Out of the 32 patients who were treated with corticosteroids at baseline in the AxiG trial (EudraCT 2011-000900-16) 17 could lower and 5 could stop their steroids during treatment with axitinib. PFS was identical for patient with or without need for steroids at baseline in the AxiG trial but OS was numerically superior for patients not in need for steroids at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis:

   * Histologically confirmed diagnosis of World Health Organization Grade IV malignant glioma (glioblastoma or gliosarcoma);
   * Documentation of recurrent (or progressive according to RNAO criteria) glioblastoma following prior treatment with surgery (resection or biopsy), radiation therapy and temozolomide chemotherapy;
   * A formalin-fixed, paraffin-embedded (FFPE) tumor tissue block or 15 unstained slides (10 minimum) obtained from an archival FFPE tumor tissue block will be required.
   * Presence of a measurable tumor lesion that is characterized by gadolinium enhancement on T1-MRI of the brain (with a shortest diameter of >5 mm) and enhanced lesion to normal brain uptake on FET-PET imaging of the brain;
   * If first recurrence of GBM is documented by MRI, an interval of at least 12 weeks after the end of prior radiation therapy is required unless there is either: i) histopathologic confirmation of recurrent tumor, or ii) new enhancement on MRI outside of the radiotherapy treatment field.
   * An interval of >28 days and full recovery (ie, no ongoing safety issues) from surgical resection and an interval of >4 weeks after the last administration of any other treatment for glioblastoma.
2. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative, as allowed by local guidance/practice) has been informed of all pertinent aspects of the study.
3. Patients who are willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
4. Age ≥ 18 years.
5. Estimated life expectancy of at least 3 months.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
7. No evidence of pre-existing uncontrolled hypertension as documented by 2 baseline blood pressure (BP) readings taken at least 1 hour apart. The baseline systolic BP readings must be ≤ 140 mm Hg, and the baseline diastolic BP readings must be ≤ 90 mm Hg. Use of antihypertensive medications to control BP is allowed.
8. Adequate bone marrow function, including:

   1. Absolute neutrophil count (ANC) ≥ 1,500/mm3 or ≥ 1.5 x 109/L;
   2. Platelets ≥ 100,000/mm3 or ≥ 100 x 109/L;
   3. Hemoglobin ≥ 9 g/dL (may have been transfused).
9. Adequate renal function, including:

   1. Estimated creatinine clearance ≥ 30 mL/min as calculated using the Cockcroft-Gault (CG) equation;
   2. Urinary protein <2+ by urine dipstick. If dipstick is ≥ 2+, then 24-hour urinary protein <2 g per 24 hours.
10. Adequate liver function, including:

    1. Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN);
    2. AST and ALT ≤ 2.5 x ULN.
11. Serum pregnancy test (for females of childbearing potential) negative at screening.
12. Male patients able to father children and female patients of childbearing potential and at risk for pregnancy must agree to use 2 highly effective methods of contraception throughout the study and for at least 90 days after the last dose of assigned treatment.

Exclusion criteria:

1. Any of the following prior cancer therapies:

   * Prior immunotherapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways;
   * Prior therapy with axitinib as well as any prior therapies with other VEGF pathway inhibitors (including bevacizumab).
2. Participation in other therapeutic studies within 4 weeks prior to enrollment in the current study.
3. Persisting toxicity related to prior therapy NCI CTCAE v4.03 Grade > 1; however, sensory neuropathy Grade ≤ 2 is acceptable.
4. Current or prior use of immunosuppressive medication within 7 days prior to enrollment, except for steroid treatment needed to palliate glioblastoma associated neurological symptoms and intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection);
5. No treatment with enzyme inducing anti-epileptic drugs (EIAED) during and at least 14 days before the administration of axitinib;
6. Known severe hypersensitivity reactions to monoclonal antibodies (Grade > 3), any history of anaphylaxis.
7. Known prior or suspected hypersensitivity to study drugs or any component in their formulations.
8. Diagnosis of any other malignancy within 5 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix, or low-grade (Gleason 6 or below) prostate cancer on surveillance with no plans for treatment intervention (eg, surgery, radiation or castration).
9. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agents. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
10. Gastrointestinal abnormalities including:

    * Inability to take oral medication;
    * Requirement for intravenous alimentation;
    * Prior surgical procedures affecting absorption including total gastric resection;
    * Treatment for active peptic ulcer disease in the past 6 months;
    * Active gastrointestinal bleeding, unrelated to cancer, as evidenced by clinically significant hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
    * Malabsorption syndromes.
11. Active infection requiring systemic therapy.
12. Diagnosis of prior immunodeficiency or organ transplant requiring immunosuppressive therapy, or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
13. Any test for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating acute or chronic infection.
14. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated influenza vaccines).
15. Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access device or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
16. Evidence of inadequate wound healing (including dehiscence of the craniotomy scar).
17. Grade ≥ 3 hemorrhage within 4 weeks of patient enrollment.
18. Any of the following in the previous 12 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, LVEF less than LLN, clinically significant pericardial effusion, cerebrovascular accident, transient ischemic attack.
19. Any of the following in the previous 6 months: deep vein thrombosis or symptomatic pulmonary embolism.
20. Evidence of tumor involvement of the myocardium or pericardium or tumor thrombus extending to the heart.
21. Current use or anticipated need for treatment with drugs or foods that are known strong CYP3A4/5 inhibitors, including their administration within 10 days prior to patient enrollment (eg, grapefruit juice or grapefruit/grapefruit-related citrus fruits [eg, Seville oranges, pomelos], ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil, and conivaptan). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
22. Current use or anticipated need for drugs that are known strong CYP3A4/5 inducers, including their administration with 10 days prior to patient enrollment(eg, phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, rifapentin, clevidipine, St John's wort).
23. Pregnant female patients, breastfeeding female patients.
24. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, uncontrolled asthma, and pneumonitis or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
6-month PFS% | 24 weeks
  The percentage of patients who are alive and free-from confirmed tumor progression at 6-month (24 weeks).

SECONDARY OUTCOMES:
Median OS (Overall survival) | an average of 1 year
  Estimate OS according to stratum and for the total study population by Kaplan-Meier estimates.
Objective Tumor Response (OR) | up to 24 weeks
  To assess anti-tumor activity by evaluating the OR as assessed by iRANO criteria.
Overall Safety profile | Overall safety will be continuously monitored throughout the duration of the treatment, until one month after last patient visit.
  To evaluate the overall safety profile of avelumab in combination with axitinib by evaluating the adverse events (AEs) and laboratory abnormalities as graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Evolution of neuro-cognitive function | Up to 24 weeks; on week 1, week 9 of the treatment phase and week 20 of the follow-up phase
  Document neuro-cognitive function by Cogstate computer based neurocognitive assessment during study treatment.
Continuous activity | Activity will be continuously monitored for 2 weeks, two times with an interval of 6 weeks during the treatment phase.
  Assess the activity level in treated recGB patients by continuous activity tracking during study treatment by means of an activity tracking device.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman HS, Prados MD, Wen PY, Mikkelsen T, Schiff D, Abrey LE, Yung WK, Paleologos N, Nicholas MK, Jensen R, Vredenburgh J, Huang J, Zheng M, Cloughesy T. Bevacizumab alone and in combination with irinotecan in recurrent glioblastoma. J Clin Oncol. 2009 Oct 1;27(28):4733-40. doi: 10.1200/JCO.2008.19.8721. Epub 2009 Aug 31. PMID 19720927
- [Background] Kreisl TN, Kim L, Moore K, Duic P, Royce C, Stroud I, Garren N, Mackey M, Butman JA, Camphausen K, Park J, Albert PS, Fine HA. Phase II trial of single-agent bevacizumab followed by bevacizumab plus irinotecan at tumor progression in recurrent glioblastoma. J Clin Oncol. 2009 Feb 10;27(5):740-5. doi: 10.1200/JCO.2008.16.3055. Epub 2008 Dec 29. PMID 19114704
- [Background] Lamborn KR, Yung WK, Chang SM, Wen PY, Cloughesy TF, DeAngelis LM, Robins HI, Lieberman FS, Fine HA, Fink KL, Junck L, Abrey L, Gilbert MR, Mehta M, Kuhn JG, Aldape KD, Hibberts J, Peterson PM, Prados MD; North American Brain Tumor Consortium. Progression-free survival: an important end point in evaluating therapy for recurrent high-grade gliomas. Neuro Oncol. 2008 Apr;10(2):162-70. doi: 10.1215/15228517-2007-062. Epub 2008 Mar 4. PMID 18356283
- [Background] Meyers CA, Scheibel RS. Early detection and diagnosis of neurobehavioral disorders associated with cancer and its treatment. Oncology (Williston Park). 1990 Jul;4(7):115-22; discussion 122, 126-7, 130. PMID 1697183
- [Background] Taphoorn MJ, Klein M. Cognitive deficits in adult patients with brain tumours. Lancet Neurol. 2004 Mar;3(3):159-68. doi: 10.1016/S1474-4422(04)00680-5. PMID 14980531
- [Background] Bosma I, Vos MJ, Heimans JJ, Taphoorn MJ, Aaronson NK, Postma TJ, van der Ploeg HM, Muller M, Vandertop WP, Slotman BJ, Klein M. The course of neurocognitive functioning in high-grade glioma patients. Neuro Oncol. 2007 Jan;9(1):53-62. doi: 10.1215/15228517-2006-012. Epub 2006 Oct 3. PMID 17018697
- [Background] Meyers CA, Hess KR, Yung WK, Levin VA. Cognitive function as a predictor of survival in patients with recurrent malignant glioma. J Clin Oncol. 2000 Feb;18(3):646-50. doi: 10.1200/JCO.2000.18.3.646. PMID 10653880
- [Background] Li J, Bentzen SM, Li J, Renschler M, Mehta MP. Relationship between neurocognitive function and quality of life after whole-brain radiotherapy in patients with brain metastasis. Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):64-70. doi: 10.1016/j.ijrobp.2007.09.059. PMID 18406884
- [Background] Brown PD, Jensen AW, Felten SJ, Ballman KV, Schaefer PL, Jaeckle KA, Cerhan JH, Buckner JC. Detrimental effects of tumor progression on cognitive function of patients with high-grade glioma. J Clin Oncol. 2006 Dec 1;24(34):5427-33. doi: 10.1200/JCO.2006.08.5605. PMID 17135644
- [Result] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895